CLINICAL TRIAL: NCT03955549
Title: Insight Enhancement Program vs. Metacognitive Training for Psychosis in Patients With Schizophrenia: A Three-Armed Comparative Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agiad Psychiatry Hospital (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ahmed Ahmed Dobie, Specialist of Psychiatry, Agiad Psychiatry Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-09
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Insight Enhancement Program; Insight Enhancement Therapy; Metacognitive Training for Psychosis; Psychotherapeutic Interventions for Schizophrenia; Research on Schizophrenia in Egypt
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Therapeutics; Control Groups

STUDY DESIGN:
Intervention Model Description: This will be a three-armed parallel group, assessor-blind, randomized controlled trial comparing "Insight Enhancement Program" (IEP) and "Metacognitive Training for Psychosis" (MCT) with "Treatment As Usual" (TAU). Once the participant gives his/her consent, he/she will be randomized either to (IEP+TAU), or (MCT+TAU), or (TAU). Both interventions consist of eight session administered over 4 weeks. The total study duration will be 2 months as participants must be on a fixed dose of the antipsychotic medication for 4 weeks prior to starting the interventions. Participants will be assessed twice during the study period; the first assessment will be after 4 weeks of receiving the antipsychotic medication prior to starting the interventions, and the final assessment will be at the end of the study after finishing the interventions. A total of 120 participants will be recruited in the study and randomized across the three groups in a 1:1:1 proportion.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to treatment allocation, and specific measures will be undertaken to preserve blinding and prevent a Rosenthal effect (e.g., assessors will not be employees of the same hospital, and before each assessment participants will be explicitly instructed not to disclose their group assignment to the assessor).
  Randomization will be according to a randomization plan using stratified permuted block randomization with each block containing four participants. This method will be used to achieve balance among groups in terms of subjects' baseline characteristics. Stratified randomization is achieved by generating a separate block for each covariate such as age & gender.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Insight Enhancement Program (IEP) (Experimental): The insight enhancement program is a dynamo-cognitive therapeutic modality with the main target of improving insight in psychotic patients as a means of improving their overall outcome.
  Interventions: Behavioral: Insight Enhancement Program (IEP); Drug: Treatment As Usual (TAU)
- Metacognitive Training for Psychosis (MCT) (Experimental): The metacognitive training program, developed by Moritz et al. (Moritz & Woodward, 2007) targets cognitive biases putatively involved in the formation and maintenance of psychotic symptoms.
  Interventions: Behavioral: Metacognitive Training for Psychosis (MCT); Drug: Treatment As Usual (TAU)
- Treatment As Usual (TAU) (Active Comparator): Treatment as usual will be used as a control condition to assure ethicality of our procedure.
  Medications: In order to standardize treatment, Risperidone (Risperdal ) will be used as the antipsychotic medication in all three groups with a dose up to 6-8 milligrams according to clinical severity. The same dose will be used for 1 month prior to starting interventions). In case of occurrence of mild extrapyramidal symptoms associated with high doses of risperidone, an anticholinergic drug (Benztropine) might be used.
  Interventions: Drug: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Insight Enhancement Program (IEP) — IEP is comprised of 8 sessions, administered twice weekly, across a one month period. The session duration is 60-90 minutes. IEP will be administered in a group format with 8-12 patients in each group.
  During sessions, different topics representing 8 different stages of illness are discussed according to a chronological schedule. These stages are presented on an Illness March Graph (IMG) and include: Stage I: Personality formation, Stage II: Pre onset confusion, Stage III: Prodroma, Stage IV: The illness, Stage V: Resistance, Stage VI: Remission, Stage VII: Maintenance, Stage VIII: Relapse. Patients actively participate through the exchange of their own experiences and interpretations, which are then reinterpreted by the therapist and by the patients themselves.
  Other Names: Insight Enhancement Therapy
  Arms: Insight Enhancement Program (IEP)
Behavioral: Metacognitive Training for Psychosis (MCT) — The training consists of eight modules that are administered within the framework of a group intervention program that involves eight 1-hour group sessions with 4 to 10 patients in each group. MCT is manualized and currently available in thirty languages and can been downloaded via the following web address: http://www.uke.de/mct. Among the problematic thinking styles recognized as potential contributors to the development of delusions are attributional distortions (module 1), a jumping to conclusions bias (module 2 and 7), a bias against disconfirmatory evidence (module 3), deficits in theory of mind (module 4 and 6), over-confidence in memory errors (module 5) and depressive cognitive patterns (module 8).
  Other Names: Metacognitive Training
  Arms: Metacognitive Training for Psychosis (MCT)
Drug: Treatment As Usual (TAU) — Treatment As Usual (TAU) consists of psychiatric management by a clinical team including at least one psychiatrist and one psychologist. Treatment involves antipsychotic medication, regular office-based contacts with the clinical team for treatment monitoring, recreational group activities, and unstructured psycho-educational groups. Participants in the interventional groups also will receive TAU.
  Medications: In order to standardize treatment, Risperidone (Risperdal ) will be used as the antipsychotic medication in all three groups with a dose up to 6-8 milligrams according to clinical severity. The same dose will be used for 1 month prior to starting interventions). In case of occurrence of mild extrapyramidal symptoms associated with high doses of risperidone, an anticholinergic drug (Benztropine) might be used.
  Other Names: Control Group

SUMMARY:
The aim of this study is to explore new safe effective psychotherapeutic interventions for schizophrenia through assessing the efficacy and acceptability of complementary "Insight Enhancement Program" (IEP) and "Metacognitive Training for Psychosis" (MCT), in relation to each other, and in relation to "Treatment As Usual" (TAU). It is hypothesized that at the end of therapy, compared to "Treatment As Usual", patients undergoing whether (IEP) or (MCT) will display a significant reduction in psychopathology particularly positive symptoms and delusional ideation, and a significant improvement in Insight and metacognitive capacity. Additionally, it is hypothesized that the acceptance of (IEP) and (MCT) will be higher than acceptance of (TAU). This study also aims to examine whether metacognition is associated with insight even after controlling for the effects of psychiatric symptomatology.

DETAILED DESCRIPTION:
Specific aims include:

1. Aim #1: Evaluate the efficacy of complementary "Insight Enhancement Program" (IEP), compared to TAU, in reducing psychopathology particularly positive symptoms and delusional ideation, and improving insight and metacognitive capacity as well as social functioning.
2. Aim #2: Evaluate the efficacy of complementary "Metacognitive Training for Psychosis" (MCT), compared to TAU, in reducing psychopathology particularly positive symptoms and delusional ideation, and improving insight and metacognitive capacity as well as social functioning.
3. Aim #3: Compare the efficacy of complementary "Insight Enhancement Program" (IEP), compared to "Metacognitive Training for Psychosis" (MCT), in reducing psychopathology and improving insight and metacognitive capacity as well as social functioning.
4. Aim #4: Examine the associations between insight, metacognition, and psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of a Schizophrenia Spectrum Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM5).
* A present or prior episode of delusional symptoms, as assessed via clinical interview.
* Within the first five years since the onset of psychosis.
* Age between 18 and 65 years.
* Egyptian Nationality.
* Fluent command of the Arabic language.
* Capacity to understand the study description and provide informed consent.

In order to examine the efficacy of IEP and MCT in cases with minor symptom load, no minimum symptom threshold was defined for inclusion.

Exclusion Criteria:

* Comorbid Substance Dependence Disorder.
* Comorbid medical conditions, whose pathology or treatment could alter the presentation or treatment of schizophrenia.
* Intellectual disability (IQ of less than 70).
* Known sensitivity to Risperidone.
* Pregnant or Breast feeding women.
* Scores of 5 or higher on the PANSS hostility item and of 6 or higher on PANSS suspiciousness item (As group settings can be disrupted by behavioral disturbances, patients with very severe forms of delusions, formal thought disorder and hostility should refrain from participating in MCT or IEP until some remission has taken place).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Mean Change in Psychopathology as measured by The Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The Positive and Negative Syndrome Scale for Schizophrenia (PANSS) is a 30-item, seven-point (1-7) scale and it is the most widely used instrument for the assessment of schizophrenia symptoms in clinical trials. Ratings follow semi-structured interviews and clear standard operating procedures. Symptoms are rated according to their presence in the past 2 weeks. The PANSS was used many times before in trials of MCT & insight in schizophrenia, which makes it more suitable allowing comparison of results.
Mean Change in Psychopathology as measured by The Psychotic Symptom Rating Scale (PSYRATS) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The PSYRATS is a 17-item multidimensional measure of more qualitative aspects of hallucinations and delusions. Symptoms are rated over the past 2 weeks. Two subscales exist; for auditory hallucinations (11 items), and for delusions (6 items).
Mean Change in Insight Scores as measured by The Scale to Assess Unawareness of Mental Disorder (SUMD) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The SUMD evaluates insight into various dimensions of the disease. The SUMD is a standardized scale that relies on a direct interview with the patient.
Mean Change in Insight Scores as measured by The Beck Cognitive Insight Scale (BCIS) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The BCIS is a self-report consisting of 15 statements rated on a 4-point Likert scale. It is divided into 2 subscales; self-reflectiveness, and self-certainty. Self-reflectiveness consists of 9 items measuring objectivity, reflectiveness and openness to feedback. Self-certainty consists of 6 items measuring decision-making and resistance to feedback. Overall cognitive insight was defined by Beck and associates as the difference between self-reflectiveness and self- certainty and labeled composite index.
Mean Change in Metacognition Scores as measured by The Metacognition Assessment Scale - Adapted version (MAS-A) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The MAS-A is scored on the basis of the transcript of the Indiana Psychiatric Illness Interview (IPII). Scoring is performed by a consensus group of at least three trained raters. The four domains of metacognition are reflected in the four ordinal complexity scales of the MAS-A: self-reflectivity, understanding the other's mind, decentration, and mastery. The raters assign one point for each function on each scale that they judge is accomplished in the transcript.

SECONDARY OUTCOMES:
Mean Change in Scores as measured by The Personal and social performance scale (PSP) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The PSP was used to assess subjects' social functioning. Patients' functioning is assessed in four core areas: Socially useful activities; personal and social relationships; self-care; and disturbing and aggressive behaviours. A global item is rated by the interviewer, ranging from 1 to 100 at 10-point intervals with lower scores indicating poorer functioning. The PSP shows good psychometric properties.
Mean Change in Neuropsychological Functioning Scores as measured by The Trail making test (TMT) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The Trail Making Test (TMT) Part A and B will be used to assess sustained attention, visual-spatial search, and psychomotor speed. The A-form requires the subject to combine numbers as fast as possible in ascending order. In the B-part, the subject has to combine numbers and letters as quickly as possible in both alternating and ascending fashion. The rating is based on the number of seconds needed to complete the test.
Mean Change in Neuropsychological Functioning Scores as measured by The Digit Symbol Substitution Test (DSST) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The Digit Symbol Substitution Test (DSST) is part of the Wechsler Adult Intelligence Scale (Wechsler, 2008), and is used to assess visuo-motor processing speed. The total score on this test is based on the amount of correctly completed symbols within 120 seconds.
Mean Change in Neuropsychological Functioning Scores as measured by The story subtest of the Rivermead Behavioural Memory Task. | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  This test will be administered to determine immediate and delayed recall.
Mean Change in Neuropsychological Functioning Scores as measured by The Porteus Mazes task. | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  The Porteus Mazes task was used to assess reasoning and problem solving.
Mean Change in IQ as measured by The Wechsler Adult Intelligence Scale (WAIS-III) | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  • The Wechsler Adult Intelligence Scale (WAIS) III, (Wechsler, 1997). Current IQ was measured using a short form of the Wechsler Adult Intelligence Scale (WAIS) III composed of 4 subtests: information, arithmetic, block design, and digit symbol and developed for use in schizophrenia (Blyler et al., 2000).
Mean Change in Self-Esteem Scores as measured by The Rosenberg Self-esteem Scale (RSES) - Arabic Version - | Pre-Intervention at Week 4, and Post-Intervention at Week 8
  • The 10-item Rosenberg scale is considered the gold-standard for the assessment of self-esteem, and its good validity and reliability have been confirmed for the Arabic version
Adverse Events will be measured by The Systematic Monitoring of Adverse Events Related to Treatments Checklist (SMARTS) | At Baseline, Week 2, Week 4, Week 6, Week 8
  The SMARTS checklist aims to strike a balance between brevity and capturing the most common and important antipsychotic side effects.

OTHER OUTCOMES:
Subjective Acceptance of the Interventions as measured by an Acceptance Questionnaire | At Week 8
  To assess acceptance, feasibility and subjective efficacy of the interventions, participants will be asked to anonymously appraise the training at post-treatment. The questionnaire is modeled after versions administered in previous trials (Moritz and Woodward, 2007; Moritz et al., 2011), and is comprised of ten questions posed on a five-point Likert scale (1=fully agree to 5=fully disagree). Acceptance and feasibility will also be assessed with the frequency of unattended sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Dobie, Msc., Principal Investigator — Agiad Psychiatry Hospital; Mai M. El-Bassosy, Msc., Principal Investigator — Agiad Psychiatry Hospital
Locations (1):
- Agiad Psychiatry Hospital, Ţalkhā, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
A plan is still being put together
Supporting Information: SAP, CSR
Time Frame: 6 months after publishing
Access Criteria: Other Researchers